CLINICAL TRIAL: NCT00364845
Title: A Randomised Single-Blind Study to Improve Health-related Quality of Life as Measured by the Short-Form 36 (SF-36) Vitality Score by Correcting Anemia With Aranesp (Darbepoetin Alfa) in the Elderly.
Brief Title: STIMULATE Study: Anemia Correction and Health-related Quality of Life (HRQoL) Outcomes in Elderly Chronic Kidney Disease (CKD) Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The reason for the discontinuation of the study is difficulty with recruitment and timely enrolment and is not related to safety concerns
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20050122
Record Dates: First submitted 2006-08-14; First posted 2006-08-16 (Estimated); Results first posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-04

CONDITIONS: Anemia; Chronic Kidney Disease
Keywords: Quality of Life; Chronic Kidney Disease; Anemia
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Darbepoetin alfa (Active Comparator): Single-blind darbepoetin alfa administered by subcutaneous injection (SC) every other week until hemoglobin (Hgb) was stable (2 consecutive Hgb values between 120 and 135 g/L), then every month for up to 9 months.
  Interventions: Drug: Darbepoetin alfa
- Placebo (Placebo Comparator): Single-blind placebo administered by subcutaneous injection (SC) every other week until week 16, then every month for up to 9 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darbepoetin alfa — Starting dose was calculated at 0.75 micrograms per kilogram (μg/kg) body weight at randomization, rounded to nearest prefilled syringe dose unit. Dose was titrated incrementally. Monthly dose was initially double the every 2 week dose at time of conversion.
  Other Names: Aranesp®
  Arms: Darbepoetin alfa
Drug: Placebo — Prefilled syringe placebo, to match active arm
  Arms: Placebo

SUMMARY:
Treatment of anemia associated with chronic kidney disease (CKD) during 36 weeks with safety follow up phase of 52 weeks

DETAILED DESCRIPTION:
This is a multicentre, randomised, single-blind, placebo-controlled, two-arm parallel group study assessing the effect of anaemia correction and Hb maintenance with darbepoetin alfa in elderly CKD patients for 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3-5 CKD not on dialysis
* Patients ≥ 70 years of age
* Haemoglobin < 110g/L at screening
* Transferrin saturation ≥ 15% at screening

Exclusion Criteria:

* Clinical history of type 2 diabetes mellitus
* Anticipating or scheduled to go on renal replacement therapy in the next year, including renal transplant
* Uncontrolled hypertension on two separate measurements during screening
* Use of any erythropoietic protein within 12 weeks of screening

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 21 September 2006 through 6 November 2007
Period: Overall Study
Arm/Group | Darbepoetin Alfa | Placebo
Started | 28 | 23
Completed | 17 (Completed 36-week titration/treatment phase) | 12 (Completed 36-week titration/treatment phase)
Not Completed | 11 | 11
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 8 | 8
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Darbepoetin Alfa | Placebo | Total
Number analyzed (Participants) | 28 | 23 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 79.2 (4.9) | 81.0 (5.1) | 80.0 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 15 | 14 | 29
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 26 | 22 | 48
  Asian | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Short Form 36 Health Survey Questionnaire (SF-36) Vitality Subscale Score at Week 24
Description: The SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The vitality sub-score assesses energy and fatigue, and ranges from 0 (worst) - 100 (best).
Time Frame: Week 24
Population: Subset of Full Analysis Set, composed of all randomized participants with available data.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Darbepoetin Alfa | Placebo
Number analyzed (Participants) | 19 | 18
Units on a scale | 51.4 (1.6) | 46.7 (2.8)

2. Secondary Outcome: Number of Participants With Hemoglobin (Hb) ≥ 110 g/L
Description: Number of participants achieving a Hemoglobin (Hb) value ≥ 110 g/L during the evaluation period.
Time Frame: Evaluation Period (Weeks 22-36)
Population: Subset of Full Analysis Set, composed of all randomized participants with available data
Measure: Number; unit: Participants
Arm/Group | Darbepoetin Alfa | Placebo
Number analyzed (Participants) | 20 | 18
Participants | 19 | 7
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; Proportion achieving target = 0.389, 95% CI [0.173 to 0.643]
Statistical Analysis 2: Comparison: Darbepoetin Alfa; Test type: Superiority or Other; Proportion achieving target = 0.950, 95% CI [0.751 to 0.999]

3. Secondary Outcome: Mean Hemoglobin During the Evaluation Period
Time Frame: Evaluation Period (Weeks 22-36)
Population: Subset of Full Analysis Set, composed of all randomized participants with available data
Measure: Mean (95% Confidence Interval); unit: g/L
Arm/Group | Darbepoetin Alfa | Placebo
Number analyzed (Participants) | 20 | 18
g/L | 125.85 [121.84 to 129.86] | 104.50 [99.35 to 109.65]

4. Secondary Outcome: Euroqol 5 Dimension (EQ-5D) Utility Score at Week 24
Description: The EQ-5D is a patient-completed, multidimensional measure of health related quality of life. The instrument is applicable to a wide range of health conditions and treatments and results in a single index score. The EQ-5D descriptive health profile comprises five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension comprises three levels (no problems, some/moderate problems, extreme problems). A unique EQ-5D health state is defined by combining one level from each of the five dimensions. EQ-5D index values range from -0.59 to 1.00. Higher EQ-5D Index scores represent better health status.
Time Frame: Week 24
Population: Subset of Full Analysis Set, composed of all randomized participants with available data
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Darbepoetin Alfa | Placebo
Number analyzed (Participants) | 19 | 16
Units on a scale | 0.763 [0.683 to 0.844] | 0.712 [0.598 to 0.826]

ADVERSE EVENTS:
Time Frame: Up to 46 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Darbepoetin Alfa | Placebo
Serious Adverse Events (participants affected / at risk) | 7/28 | 5/23
Other Adverse Events (participants affected / at risk) | 21/28 | 18/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa (N=28) | Placebo (N=23)
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Adrenal mass (Endocrine disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Encephalitis (Nervous system disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa (N=28) | Placebo (N=23)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 1 | 3
Fatigue (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 2
C-reactive protein increased (Investigations) | 2 | 0
Gout (Metabolism and nutrition disorders) | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Dizziness (Nervous system disorders) | 3 | 4
Headache (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 2 | 3
Paraesthesia (Nervous system disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.